CLINICAL TRIAL: NCT05161832
Title: Impact of Kinesiophobia on Descending Corticospinal and Bulbospinal Projections During Experimental Pain : A Randomised Controlled Trial
Brief Title: Impact of Kinesiophobia on Descending Corticospinal and Bulbospinal Projections
Acronym: EchoKinésio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Guillaume Léonard, Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2022-4356
Record Dates: First submitted 2021-11-26; First posted 2021-12-17 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Kinesiophobia
Keywords: kinesiophobia; experimental pain; corticospinal excitability; conditioned pain modulation; input output curves
MeSH Terms: conditions — Kinesiophobia | interventions — Nocebo Effect

STUDY DESIGN:
Intervention Model Description: Participants will attend two experimental sessions at the Research Center on Aging of the Centre Intégré Universitaire de Santé et de Services Sociaux de l'Estrie, Sherbrooke. During the first one, the efficacy of their excitatory and inhibitory mechanisms will be assessed (thermode and cold water bath) and during the second one, their corticospinal excitability will be assessed by transcranial magnetic stimulation (before and during induced pain + placebo or nocebo echography of shoulder). Subjects will be randomized between 2 arms, nocebo (bad fake result) or placebo echography (good fake result). Participants will be allocated using minimization with 2 factors (age and sex). The two sessions will be separated by at least 48 hours.
Who Masked: Participant, Investigator
Masking Description: The principal investigators will be blinded by anonymization of the subjects and will not be present during the ultrasound. Participants will be notified of their group allocation at the end of their experimental session (after the experiment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nocebo (Experimental): Ultrasound with fake results of rotator cuff injury.
  Interventions: Behavioral: Nocebo
- placebo (Active Comparator): Ultrasound with fake results of the healthy rotator cuff.
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Nocebo — Nocebo ultrasound with diagnosis of a fake shoulder cuff injury.
  Arms: nocebo
Behavioral: Placebo — Placebo ultrasound with no diagnosis of injury.
  Arms: placebo

SUMMARY:
Fear of movement (kinesiophobia) is a phenomenon commonly observed in people suffering from chronic pain. The aims of this project are to better understand the neurophysiological basis of this phenomenon, in particular 1) the effect of kinesiophobia (induced by nocebo intervention) on the excitability of corticospinal projections and 2) the association between kinesiophobia and top-down inhibitory mechanisms.

DETAILED DESCRIPTION:
The study will include 44 healthy (pain-free) participants. Corticospinal measurements will be taken before and after the application of capsaicin cream (experimental pain paradigm). The investigators will manipulate kinesiophobia levels (assessed using the Tampa Kinesiophobia Scale) upward by pretending to diagnose a musculoskeletal problem in half of the participants (nocebo ultrasound), and will measure the efficacy of top-down inhibitory mechanisms using a counter-irritation paradigm (thermode and cold pressor test : the subjects will be subjected to 5 thermal stimulations, 7 mechanical stimulations and 1 water bath at 10°C of the hand) and corticospinal parameters using transcranial magnetic stimulation.

Together, these results will allow a better understanding of the mechanisms associated with a predictor of pain onset (such as kinesiophobia), by studying its interactions with endogenous pain inhibition systems and the motor system, in order to develop relevant prophylactic treatments.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old or older
* Healthy Volunteers
* Capable of understanding instructions
* Abstain from tobacco and caffeine 2 hours before data collection
* Abstain from short-acting analgesics 6 hours before data collection

Exclusion Criteria:

* A painful condition or chronic pain
* Neurological disorders
* Shoulder pathology
* Skin diseases
* Capsaicin allergy
* Raynaud's syndrome
* Epilepsy
* Intracranial metallic foreign bodies, hearing aids and cochlear implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-07-29 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Corticospinal excitability | 1 hour
  The corticospinal excitability will be assessed using motor evoked potentials at different intensity of stimulation (from motor threshold to maximal amplitude response).

SECONDARY OUTCOMES:
downward inhibition of pain | 1 hour
  Inhibitory mechanisms will be assessed by comparing pain levels (measured using a computerized visual analog scale [0 = no pain; 10 = worst pain imaginable]) evoked by a test stimulus before and after a conditioning stimulus.
  Pain levels evoked by the test stimulus before the conditioning stimulus will be subtracted from pain levels evoked by the test stimulus after the pain stimulus, such that a positive score represents increased pain (hyperalgesia) and a negative score represents decreased pain (hypoalgesia, i.e., inhibitory mechanisms).

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Leonard, Pr, Study Director — Université de Sherbrooke
Locations (1):
- Centre de Recherche sur le Vieillissement, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No